CLINICAL TRIAL: NCT00450619
Title: A Randomized Phase 2.5 Study of (153)Sm-EDTMP (Quadramet) With or Without a PSA/TRICOM Vaccine in Men With Androgen-Insensitive Metastatic Prostate Cancer
Brief Title: 153Sm-EDTMP With or Without a PSA/TRICOM Vaccine To Treat Men With Androgen-Insensitive Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Gulley, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 070106; 07-C-0106
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Results first posted 2013-07-01 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Prostate Cancer
Keywords: Radionuclide; Immunotherapy; Radiation; PSA; Hormone Refractory Prostate Cancer; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — samarium Sm-153 lexidronam; sargramostim; rV-Tricom

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A -EDTMP Alone (Experimental): Patients receive samarium Sm 153 lexidronam pentasodium 1 mCi/Kg intravenous (IV) over 1 minute on day 8. Treatment repeats every 12 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Samarium Sm 153 lexidronam pentasodium
- Arm B - 153SmEDTMP with vaccine (Experimental): Patients receive recombinant vaccinia-TRICOM vaccine 2 x 10^8 PFU subcutaneously (SC) on day 1. Patients also receive recombinant fowlpox-TRICOM vaccine 1 x 10^9 PFU SC on days 15 and 29 and sargramostim (GM-CSF)100 mcg/injection SC x 4 days. Treatment with recombinant fowlpox-TRICOM vaccine and GM-CSF* repeats every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive samarium Sm 153 lexidronam pentasodium 1 mCi/Kg as in arm I.
  Interventions: Radiation: Samarium Sm 153 lexidronam pentasodium; Biological: Sargramostim; Biological: Recombinant vaccinia-TRICOM vaccine; Biological: Recombinant fowlpox-TRICOM vaccine

INTERVENTIONS:
Radiation: Samarium Sm 153 lexidronam pentasodium — 1 mCi/Kg given intravenous (IV)over 1 minute on day 8.
Biological: Sargramostim — 100 mcg/injection x 4 days given subcutaneously
  Arms: Arm B - 153SmEDTMP with vaccine
Biological: Recombinant vaccinia-TRICOM vaccine — 2 x 10^8 PFU given subcutaneously on day 1.
  Arms: Arm B - 153SmEDTMP with vaccine
Biological: Recombinant fowlpox-TRICOM vaccine — 1 x 10^9 PFU given subcutaneously on days 15 and 29
  Arms: Arm B - 153SmEDTMP with vaccine

SUMMARY:
Background:

* No treatment is known to improve survival for prostate cancer patients who have not been helped by previous treatments with hormones and chemotherapy.
* An experimental vaccine called prostate specific antigen (PSA)/TRICOM contains genes for a protein produced by prostate cancer cells called prostate-specific antigen (PSA). The vaccine can trigger the immune system to make cells that may be able to recognize and attack the cancer cells that make PSA.
* Granulocyte macrophage colony stimulating factor (GM-CSF) is an approved drug that is usually given to increase a patient's white blood cell count or to stimulate the immune system.
* 1Samarium-153-ethylene diamine tetramethylene phosphonate (53Sm-EDTMP) is a radioactive drug that has been approved for many years to treat advanced prostate cancer. It is given through a vein and can be targeted directly to tumors in the bone where it can relieve pain caused by bone lesions. Radiation also increases the level of certain proteins inside the tumor, making it easier for the immune system to find and kill the tumor cells.
* When laboratory mice were given just vaccine, just radiation, or a combination of both, the combination was most effective in treating tumors.

Objectives:

-To determine if combined treatment with PSA/TRICOM vaccine and 153Sm-EDTMP radiation can delay progression of prostate cancer better than radiation alone.

Eligibility:

-Patients who have advanced prostate cancer that has worsened despite treatments with hormones, have two or more bone lesions related to their prostate cancer, and have had prior treatment with docetaxel chemotherapy.

Design:

* Patients are randomly assigned to receive radiation alone (Arm A) or radiation with vaccine and sargramostim (Arm B).
* Arm A receives 153Sm-EDTMP radiation starting on study day 8 and repeated every 12 weeks.
* Arm B receives a priming vaccine on study day 1 and radiation on day 8. Radiation therapy is repeated every 12 weeks. Boosting vaccines are given on days 15 and 29 and then monthly. GM-CSF is given with each vaccination (on the day of the vaccination and for the next 3 days) to enhance the immune response. Vaccinations and GM-CSF are given as injections under the skin, usually in the thigh. Radiation therapy is given through a vein.
* Patients are monitored regularly with physical examinations, blood and urine tests, and scans to evaluate safety and treatment response.
* Patients who are human leukocyte antigen serotype within HLA-A A serotype group (HLA-A2)-positive undergo apheresis, a procedure similar to donating blood, for obtaining immune cells called lymphocytes to measure the immune response to the vaccine.

DETAILED DESCRIPTION:
Background

* There are no standard therapy options shown to prolong survival for patients with progressive disease on first-line docetaxel-based regimens for men with metastatic castration resistant prostate cancer (CRPC).
* Ninety percent of men in this population have bone metastasis.
* PSA/TRICOM vaccines as single agents can induce generation of PSA-specific T cells in the majority of patients and objective responses and PSA declines in a minority of patients. Furthermore, the generation of at least a 6-fold increase in PSA-specific T cells was significantly correlated with evidence of clinical benefit.
* Radiation can alter the phenotype of tumor cells (increase Fas, increase major histocompatibility complex (MHC), increase tumor-associated molecules and increase ICAM), making them much more amenable to immune-mediated killing.
* (153)Sm EDTMP is a beta emitter (with some gamma emissions) that targets osteoblastic bone lesions (such as those found in prostate cancer).
* (153)Sm EDTMP, at Food And Drug Administration (FDA)-approved doses used clinically for palliation of prostate cancer, can cause phenotypic changes in tumor cells, leading to improved killing of those cells in a cytotoxic T-cell assay in vitro.
* The combination of vaccine and radiation greatly increases antitumor efficacy in a murine subcutaneous tumor model.

Objectives

* Primary-A comparison of progression-free survival at 4 months between Arm A (153)Sm EDTMP alone) and Arm B (153Sm EDTMP with vaccine).
* Secondary-Objective responses, PSA outcomes, immunologic responses, toxicity, palliation and overall survival.

Eligibility

* Patients with metastatic CRPC who have 2 or more bone lesions consistent with prostate cancer and who have been treated with a docetaxel-based regimen.
* Patients with symptomatic soft tissue disease or parenchymal disease will be excluded.

Design

* Randomized phase 2.5 study.
* Sixty-eight patients to be enrolled and randomized to:

  * Arm A: (153)Sm-EDTMP: 1 mCi/kg intravenous (IV) over one minute on day 8. (153)Sm-EDTMP will be repeated every 12 weeks if there is adequate hematologic recovery.

Arm B: PROSTAC-V/TRICOM (vaccinia) 2 x 10^8 plaque forming unit (pfu) subcutaneously on day 1.

* (153)Sm-EDTMP: 1 mCi/kg IV over one minute on day 8. (153)Sm-EDTMP will be repeated every 12 weeks if there is adequate hematologic recovery. PROSTVAC-F/TRICOM (fowlpox) 1 x 10^9 pfu subcutaneously on days 15, 29, and then every 4 weeks.

ELIGIBILITY:
* INCLUSION CRITERIA:

A. Histopathological documentation of prostate cancer confirmed in the Laboratory of Pathology at the National Institutes of Health (NIH) Clinical Center, National Institutes of Health (NIH), the National Naval Medical Center, or Walter Reed Army Medical Center; or participating Institute's Department of Pathology prior to starting this study. If no pathologic specimen is available, patients may enroll with a pathologist's report showing a histologic diagnosis of prostate cancer and a clinical course consistent with the disease.

B. Must have metastatic castration resistant prostate cancer (CRPC) with at least 2 bone lesions consistent with prostate cancer metastasis and progressive disease (2 rising PSA values separated by at least one week, new or enlarging lesions consistent with prostate cancer, or clinical progression) on docetaxel for metastatic prostate cancer or inability to tolerate docetaxel.

C. Life expectancy greater than or equal to 6 months.

D. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.

E. No systemic steroid or steroid eye drop use within 2 weeks prior to initiation of experimental therapy.

F. Hematological eligibility parameters (within 16 days of starting therapy).

* Granulocyte count greater than or equal to 1,500/mm^3
* Platelet (PLT) count greater than or equal to 100,000/mm^3
* Hemoglobin (Hgb) greater than or equal to 10 Gm/dL (Transfusion may be given to accomplish this)

G. Biochemical eligibility parameters (within 16 days of starting therapy)

-Hepatic function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 times upper limit of normal; bilirubin less than 1.5 mg/dL OR in patients with Gilbert's syndrome, a total bilirubin less than or equal to 3.0 mg/dL.

H. No other active malignancies within the past 12 months (with the exception of nonmelanoma skin cancers or carcinoma in situ of the bladder and treated with curative intent) or life-threatening illnesses.

I. Willing to travel to the National Institutes of Health (NIH) or participating Institute for follow-up visits.

J. 18 years of age or greater.

K. Able to understand and sign informed consent.

L. Agree to use adequate contraception prior to study entry and for at least 4 months following the last vaccine injection.

M. Patients must remain on medical castration therapy with testosterone-suppressing therapy (e.g., gonadotropin releasing hormone (GnRH) agonist), unless they have had surgical castration.

N. Patients must have recovered from acute toxicities related to prior therapy or surgery. For chemotherapy, typically this is 3 to 4 weeks.

O. Patients who are incontinent of urine should be willing to undergo bladder catheterization to minimize the risk of radioactive contamination of clothing, bed linen, and the patient's environment.

P. Concurrent treatment with bisphosphonates is allowed. If bisphosphonates have been given within 2 weeks prior to planned (153)Sm-EDTMP, then a 99Tc whole-body scintigraphy (bone scan) will be performed to confirm uptake into lesions. Bisphosphonates will not be given within 48 hours after (153)Sm-EDTMP administration.

Q. Serum creatinine less than or equal to 1.5 times upper limit of normal OR creatinine clearance on a 24-h urine collection of greater than or equal to 60 mL/min.

EXCLUSION CRITERIA:

A. Patients should have no evidence, as listed below, of being immunocompromised:

* Human immunodeficiency virus (HIV) positivity due to the potential for decreased tolerance and risk for severe side effects.
* Hepatitis B or C positivity.
* Concurrent use of topical steroids (including steroid eye drops) or systemic steroids. This is to avoid immunosuppression which may lead to potential complications with vaccinia (priming vaccination). Nasal or inhaled steroid use is permitted.

B. Patients should have no autoimmune diseases that have required treatment, such as Addison's disease, Hashimoto's thyroiditis, systemic lupus erythematosus, Sjogren's syndrome, scleroderma, myasthenia gravis, Goodpasture's syndrome, or active Grave's disease. Patients with a history of autoimmunity that has not required systemic immunosuppressive therapy or does not threaten vital organ function, including central nervous system (CNS), heart, lungs, kidneys, skin, and gastrointestinal tract (GI) tract, will be allowed.

C. History of allergy or untoward reaction to prior vaccination with vaccinia virus or to any component of the vaccinia vaccine regimen. Note: prior vaccination with vaccinia is not required.

D. Do not administer the recombinant vaccinia vaccine if the recipient or, for at least 3 weeks after vaccination, their close household contacts (close household contacts are those who share housing or have close physical contact), are persons with active or a history of eczema or other eczematoid skin disorders; those with other acute, chronic or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds) until condition resolves; pregnant or nursing women; children 3 years of age and under; and immunodeficient or immunosuppressed persons (by disease or therapy), including HIV infection.

E. Serious intercurrent medical illness (e.g., one that requires treatment) which would interfere with the ability of the patient to carry out the treatment program, including, but not limited to, inflammatory bowel disease, Crohn's disease, ulcerative colitis, or active diverticulitis.

F. Patients with a history of cardiomyopathy or symptomatic congestive heart failure (unless stable on treatment), symptomatic arrhythmia not controlled by medication. Unstable atherosclerotic heart disease (e.g. unstable angina) who require active intervention and history of myocardial infarction or embolic stroke within the past 6 months.

G. Patients with cardiac disease who have fatigue, palpitation, dyspnea or angina with ordinary physical activity (New York Heart Association class 2 or greater) are not eligible.

H. Patients with a history of congestive heart failure or who have objective evidence of congestive heart failure by physical exam or imaging are not eligible, unless the underlying cause has been treated and patient has documented normal ejection fraction.

I. Patients with pulmonary disease who have fatigue or dyspnea with ordinary physical activity are not eligible.

J. Concurrent chemotherapy.

K. No brain metastasis or history of seizures, encephalitis, or multiple sclerosis.

L. Serious hypersensitivity reaction to egg products.

M. Prior splenectomy.

N. Contraindicated in patients who have known hypersensitivity to EDTMP or similar phosphonate compounds.

O. Patients with symptomatic soft tissue disease or parenchymal disease will be excluded.

P. Radiation therapy to bone within 4 weeks of study entry.

Q. Patients previously treated with (153)Sm-EDTMP will be excluded.

R. Patients requiring urgent local radiotherapy or orthopedic stabilization.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Cancer Institute of New Jersey, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turner JH, Claringbold PG. A phase II study of treatment of painful multifocal skeletal metastases with single and repeated dose samarium-153 ethylenediaminetetramethylene phosphonate. Eur J Cancer. 1991;27(9):1084-6. doi: 10.1016/0277-5379(91)90297-q. PMID 1720321
- [Background] Simon RM, Steinberg SM, Hamilton M, Hildesheim A, Khleif S, Kwak LW, Mackall CL, Schlom J, Topalian SL, Berzofsky JA. Clinical trial designs for the early clinical development of therapeutic cancer vaccines. J Clin Oncol. 2001 Mar 15;19(6):1848-54. doi: 10.1200/JCO.2001.19.6.1848. PMID 11251017
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Result] Christopher Ryan Heery, Ravi A. Madan, Marijo Bilusic, Joseph W. Kim, Nishith K. Singh, Myrna Rauckhorst, Clara Chen, William L. Dahut, Walter Michael Stadler, Robert S. DiPaola, Mark N. Stein, James W. Hodge, Jeffrey Schlom, James L. Gulley; Interim analysis of a phase II randomized clinical trial of samrium-153 (Sm-153) with or without PSA-TRICOM vaccine in metastatic castration-resistant prostate cancer after docetaxel. J Clin Oncol 30, 2012 (suppl; abstr 2526)
- [Result] Heery CR, Madan RA, Stein MN, Stadler WM, Di Paola RS, Rauckhorst M, Steinberg SM, Marte JL, Chen CC, Grenga I, Donahue RN, Jochems C, Dahut WL, Schlom J, Gulley JL. Samarium-153-EDTMP (Quadramet(R)) with or without vaccine in metastatic castration-resistant prostate cancer: A randomized Phase 2 trial. Oncotarget. 2016 Oct 18;7(42):69014-69023. doi: 10.18632/oncotarget.10883. PMID 27486817
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-C-0106.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A- EDTMP Alone: Patients receive samarium Sm 153 lexidronam pentasodium 1 mCi/Kg intravenous (IV) over 1 minute on day 8. Treatment repeats every 12 weeks in the absence of disease progression or unacceptable toxicity.
- Arm B - 153Sm-EDTMP With Vaccine: Patients receive recombinant vaccinia-TRICOM vaccine 2 x 10^8 PFU subcutaneously (SC) on day 1. Patients also receive recombinant fowlpox-TRICOM vaccine 1 x 10^9 PFU SC on days 15 and 29 and sargramostim (GM-CSF) 100 mcg/injection SC x 4 days. Treatment with recombinant fowlpox-TRICOM vaccine and GM-CSF* repeats every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive samarium Sm 153 lexidronam pentasodium 1 mCi/Kg as in arm I.
Period: Overall Study
Arm/Group | Arm A- EDTMP Alone | Arm B - 153Sm-EDTMP With Vaccine
Started | 22 | 22
Completed | 18 | 21
Not Completed | 4 | 1
Not completed — refused treatment after randomization | 2 | 0
Not completed — did not progress; refused further trmt | 1 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm B - 153SmEDTMP With Vaccine: Patients receive recombinant vaccinia-TRICOM vaccine 2 x 10^8 PFU subcutaneously (SC) on day 1. Patients also receive recombinant fowlpox-TRICOM vaccine 1 x 10^9 PFU SC on days 15 and 29 and sargramostim (GM-CSF) 100 mcg/injection SC x 4 days. Treatment with recombinant fowlpox-TRICOM vaccine and GM-CSF* repeats every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive samarium Sm 153 lexidronam pentasodium 1 mCi/Kg as in arm I.
- Total: Total of all reporting groups
Arm/Group | Arm A -EDTMP Alone | Arm B - 153SmEDTMP With Vaccine | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 4 | 15
  >=65 years | 11 | 18 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.73 (7.91) | 69.65 (8.5) | 67.18 (8.49)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 22 | 22 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 22 | 20 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 18 | 17 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44
Subjects requiring narcotic pain control [Number; unit: participants] | 11 | 8 | 19
Gleason Score [Median (Full Range); unit: Scores on a scale] — Gleason score is a commonly used pathology score. The range of the score is 2 to 10 with two being associated with better outcomes and 10 being associated with worse outcomes.
  Scores on a scale | 8 [6 to 9] | 7.5 [5 to 10] | 7.75 [5.5 to 9.5]
Prostate-Specific Antigen on Study [Median (Full Range); unit: ng/mL of blood] | 259.1 [22.2 to 1856] | 313.5 [4.9 to 4708] | 286.3 [13.55 to 3282]
Eastern Cooperative Oncology Group (ECOG) Performance Status [Median (Full Range); unit: Scores on a scale] — ECOG Performance Status Scale:Grade 0 - Normal activity, Fully active, able to carry on all pre-disease performance without restriction.; Grade 1 -Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., office work).; Grade 2 - In bed<50% of the time. Ambulatory and capable of all self-care.; Grade 3 - In bed >50% of the time. Capable of only limited self-care, confined to bed or chair>50% of waking hours.; Grade 4 - 100% bedridden, Completely disabled. Cannot carry on any self-care.; Grade 5 - Dead.
  Scores on a scale | 1 [0 to 1] | 1 [0 to 2] | 1 [0 to 2]
Median Days since Prior Chemotherapy [Median (Full Range); unit: Days] | 57.5 [11 to 301] | 86.5 [21 to 818] | 72 [16 to 559.5]
Lactate Dehydrogenase (serum) [Median (Full Range); unit: U/L] | 254.5 [175 to 353] | 200 [115 to 962] | 227.25 [145 to 657.5]
Hemoglobin [Median (Full Range); unit: g/dl] | 11.2 [8.8 to 13.2] | 11.1 [7.0 to 14.8] | 11.15 [7.9 to 14]
Alkaline Phosphatase [Median (Full Range); unit: U/L] | 177 [90 to 725] | 121.5 [52 to 661] | 149.25 [71 to 693]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Stable Disease at 4 Months.
Description: Response is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Stable disease is neither sufficient shrinkage to qualify for partial response (PR) nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum longest diameter (LD) since the treatment started. Partial response (PR) is at least a 30% increase in the sum of the LD of target lesions, taking as reference the baseline sum LD. Progressive Disease (PD) is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions on computed tomography (CT) or two or more lesions on bone scan.
Time Frame: 4.7 months
Measure: Number; unit: participants
Groups:
- Arm A - EDTMP Alone: Patients receive samarium Sm 153 lexidronam pentasodium 1 mCi/Kg intravenous (IV) over 1 minute on day 8. Treatment repeats every 12 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A - EDTMP Alone | Arm B - 153Sm-EDTMP With Vaccine
Number analyzed (Participants) | 18 | 21
participants | 2 | 5

2. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time to progress or die after the start of the therapy.
Time Frame: 4 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - EDTMP Alone | Arm B - 153Sm-EDTMP With Vaccine
Number analyzed (Participants) | 18 | 21
months | 1.7 [1.3 to 2.3] | 3.7 [2.4 to 4.7]
Statistical Analysis 1: Comparison: Arm A - EDTMP Alone vs Arm B - 153Sm-EDTMP With Vaccine; Test type: Superiority or Other; p = 0.041, Log Rank; Hazard Ratio (HR) = 0.5019
Statistical Analysis 2: Comparison: Arm A - EDTMP Alone vs Arm B - 153Sm-EDTMP With Vaccine; Test type: Superiority or Other; p = 0.046, Hazard Ratio; Hazard Ratio (HR) = 0.5019

3. Secondary Outcome: Toxicity
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 5 years, 5 months
Measure: Number; unit: Participants
Arm/Group | Arm A - EDTMP Alone | Arm B - 153Sm-EDTMP With Vaccine
Number analyzed (Participants) | 21 | 22
Participants | 19 | 22

4. Secondary Outcome: Number of Participants With Prostate-Specific Antigen (PSA) ≥ 30%
Description: PSA is defined by the PSA Working Group criteria. A minimum PSA decline of at least 50% must be confirmed by a second PSA value 4 or more weeks later.
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Arm A - EDTMP Alone | Arm B - 153Sm-EDTMP With Vaccine
Number analyzed (Participants) | 18 | 21
participants | 0 | 4

5. Secondary Outcome: Number of Participants With Prostate-Specific Antigen (PSA) ≥50%
Description: as for outcome 4
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Arm A - EDTMP Alone | Arm B - 153Sm-EDTMP With Vaccine
Number analyzed (Participants) | 18 | 21
participants | 0 | 3

6. Secondary Outcome: Overall Survival
Description: Time from treatment start date until date of death or date last known alive.
Time Frame: From date of randomization until death or last follow up, whichever comes first, assessed up to 14 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - EDTMP Alone | Arm B - 153Sm-EDTMP With Vaccine
Number analyzed (Participants) | 18 | 21
Months | 8.1 [3.5 to 13.3] | 9.2 [5.0 to 12.6]
Statistical Analysis 1: Comparison: Arm A - EDTMP Alone vs Arm B - 153Sm-EDTMP With Vaccine; Test type: Superiority or Other; p = 0.30, Kaplan Meier; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.37 to 1.35]

7. Secondary Outcome: Arm A: Prostate-Specific Antigen (PSA) T-cell Responses Post-vs. Pre-treatment
Description: PSA T-cell responses were measured by fluorescence activated cell sorting (FACS)-based assay for T-cells expressing type I cytokines interferon (IFN-ϓ), interleukin 2 (IL2), tumor necrosis factor alpha (TNF-a) and/or lysosome-associated membrane protein (CD107a).
Time Frame: Approximately 60 days
Population: (a)Cytokine or CD107a in CD4 or CD8. *Pts displayed pre-existing PSA-specific T-cell responses. Numbers 274, 630, and 1427 are those positive post- vs. pre-vaccination. Absolute # CD4 or CD8 producing cytokine/CD107a+/1x10(6) cells plated at start of in vitro stimulation.
Measure: Number; unit: Absolute # CD4 or CD8 producing cytokine
Arm/Group | Arm A - EDTMP Alone
Number analyzed (Participants) | 8
Absolute # CD4 or CD8 producing cytokine
  PT 11 (CD4) CD107a | 0
  PT 11 (CD4) IFN-ϓ | 0
  PT 11(CD4) IL2 | 0
  PT 11 (CD4) TNF | 0
  PT 11 (CD8) CD107a | 0
  PT 11 (CD8) IFN-ϓ | 0
  PT 11 (CD8) IL2 | 56
  PT 11 (CD8) TNF | 186
  PT 13* (CD4) CD107a | 0
  PT 13* (CD4) IFN-ϓ | 0
  PT 13* (CD4) IL2 | 0
  PT 13* (CD4) TNF | 0
  PT 13* (CD8) CD107a | 0
  PT 13* (CD8) IFN-ϓ | 0
  PT 13* (CD8) IL2 | 0
  PT 13* (CD8) TNF | 3
  PT 20* (CD4) CD107a | 0
  PT 20* (CD4) IFN-ϓ | 0
  PT 20* (CD4) IL2 | 0
  PT 20* (CD4) TNF | 0
  PT 20* (CD8) CD107a | 0
  PT 20* (CD8) IFN-ϓ | 0
  PT 20* (CD8) IL2 | 0
  PT 20* (CD8) TNF | 0
  PT 22 (CD4) CD107a | 154
  PT 22 (CD4) IFN-ϓ | 0
  PT 22 (CD4) IL2 | 0
  PT 22 (CD4) TNF | 0
  PT 22 (CD8) CD107a | 1427
  PT 22 (CD8) IFN-ϓ | 0
  PT 22 (CD8) IL2 | 0
  PT 22 (CD8) TNF | 274
  PT 25 (CD4) CD107a | 146
  PT 25 (CD4) IFN-ϓ | 0
  PT 25 (CD4) IL2 | 0
  PT 25 (CD4) TNF | 0
  PT 25 (CD8) CD107a | 0
  PT 25 (CD8) IFN-ϓ | 248
  PT 25 (CD8) IL2 | 30
  PT 25 (CD8) TNF | 630
  PT 3 (CD4) CD107a | 0
  PT 3 (CD4) IFN-ϓ | 0
  PT 3 (CD4) IL2 | 0
  PT 3 (CD4) TNF | 0
  PT 3 (CD8) CD107a | 0
  PT 3 (CD8) IFN-ϓ | 0
  PT 3 (CD8) IL2 | 14
  PT 3 (CD8) TNF | 0
  PT 5 (CD4) CD107a | 0
  PT 5 (CD4) IFN-ϓ | 0
  PT 5 (CD4) IL2 | 0
  PT 5 (CD4) TNF | 0
  PT 5 (CD8) CD107a | 0
  PT 5 (CD8) IFN-ϓ | 0
  PT 5 (CD8) IL2 | 0
  PT 5 (CD8)TNF | 25
  PT 10 (CD4) CD107a | 0
  PT 10 (CD4) IFN-ϓ | 6
  PT 10 (CD4) IL2 | 0
  PT 10 (CD4) TNF | 0
  PT 10 (CD8) CD107a | 0
  PT 10 (CD8) IFN-ϓ | 21
  PT 10 (CD8) IL2 | 0
  PT 10 (CD8) TNF | 0

8. Secondary Outcome: Arm B: Prostate-Specific Antigen (PSA) T-cell Responses Post-vs. Pre-treatment
Description: as for outcome 7
Time Frame: Approximately 60 days
Population: (a)Cytokine or CD107a in CD4 or CD8. *Pts displayed pre-existing PSA-specific T-cell responses. Numbers 786, 374, 345, 402, 821, 815, 5269, 453, 633, 1242 & 0 for PT 2 CD4/CD8 IL2 & 0 for PT 16 TNF are those positive post- vs. pre-vaccination. Absolute # CD4 or CD8 producing cytokine/CD107a+/1x10(6) cells plated at start of in vitro stimulation.
Measure: Number; unit: Absolute # CD4 or CD8 producing cytokine
Arm/Group | Arm B - 153Sm-EDTMP With Vaccine
Number analyzed (Participants) | 10
Absolute # CD4 or CD8 producing cytokine
  PT 2 (CD4) CD107a | 0
  PT 2 (CD4) IFN-ϓ | 786
  PT 2 (CD4) IL2 | 0
  PT 2 (CD4) TNF | 374
  PT 2 (CD8) CD107a | 5269
  PT 2 (CD8) IFN-ϓ | 453
  PT 2 (CD8) IL2 | 0
  PT 2 (CD8) TNF | 323
  PT 8 (CD4) CD107a | 58
  PT 8 (CD4) IFN-ϓ | 345
  PT 8 (CD4) IL2 | 0
  PT 8 (CD4) TNF | 245
  PT 8 (CD8) CD107a | 633
  PT 8 (CD8) IFN-ϓ | 136
  PT 8 (CD8) IL2 | 0
  PT 8 (CD8) TNF | 35
  PT 12 (CD4) CD107a | 0
  PT 12 (CD4) IFN-ϓ | 0
  PT 12 (CD4) IL2 | 0
  PT 12 (CD4) TNF | 0
  PT 12 (CD8) CD107a | 58
  PT 12 (CD8) IFN-ϓ | 0
  PT 12 (CD8) IL2 | 0
  PT 12 (CD8) TNF | 0
  PT 18 (CD4) CD107a | 0
  PT 18 (CD4) IFN-ϓ | 0
  PT 18 (CD4) IL2 | 75
  PT 18 (CD4) TNF | 402
  PT 18 (CD8) CD107a | 0
  PT 18 (CD8) IFN-ϓ | 0
  PT 18 (CD8) IL2 | 0
  PT 18 (CD8) TNF | 35
  PT 21 (CD4) CD107a | 0
  PT 21 (CD4) IFN-ϓ | 45
  PT 21 (CD4) IL2 | 0
  PT 21 (CD4) TNF | 0
  PT 11 (CD8) CD107a | 0
  PT 21 (CD8) IFN-ϓ | 214
  PT 21 (CD8) IL2 | 0
  PT 21 (CD8) TNF | 0
  PT 24* (CD4) CD107a | 0
  PT 24* (CD4) IFN-ϓ | 0
  PT 24* (CD4) IL2 | 149
  PT 24* (CD4) TNF | 181
  PT 24* (CD8) CD107a | 1242
  PT 24* (CD8) IFN-ϓ | 0
  PT 24* (CD8) IL2 | 8
  PT 24* (CD8) TNF | 179
  PT 14 (CD4) CD107a | 821
  PT 14 (CD4) IFN-ϓ | 0
  PT 14 (CD4) IL2 | 0
  PT 14 (CD4) TNF | 0
  PT 14 (CD8) CD107a | 0
  PT 14 (CD8) IFN-ϓ | 0
  PT 14 (CD8) IL2 | 0
  PT 14 (CD8) TNF | 0
  PT 16 (CD4) CD107a | 0
  PT 16 (CD4) IFN-ϓ | 0
  PT 16 (CD4) IL2 | 0
  PT 16 (CD4) TNF | 0
  PT 16 (CD8) CD107a | 0
  PT 16 (CD8) IFN-ϓ | 0
  PT 16 (CD8) IL2 | 9
  PT 16 (CD8) TNF | 0
  PT 26 (CD4) CD107a | 815
  PT 26 (CD4) IFN-ϓ | 0
  PT 26 (CD4) IL2 | 0
  PT 26 (CD4) TNF | 0
  PT 26 (CD8) CD107a | 149
  PT 26 (CD8) IFN-ϓ | 0
  PT 26 (CD8) IL2 | 0
  PT 26 (CD8) TNF | 0
  PT 27* (CD4) CD107a | 0
  PT 27* (CD4) IFN-ϓ | 0
  PT 27* (CD4) IL2 | 0
  PT 27* (CD4) TNF | 0
  PT 27* (CD8) CD107a | 0
  PT 27* (CD8) IFN-ϓ | 0
  PT 27* (CD8) IL2 | 0
  PT 27* (CD8) TNF | 0

9. Secondary Outcome: Objective Response (Complete Response + Partial Response)
Description: Objective response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is the disappearance of all target lesions. Partial response (PR) is at least a 30% increase in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: 4 weeks
Population: Not all participants was measureable by RECIST.
Measure: Number; unit: participants
Arm/Group | Arm A - EDTMP Alone | Arm B - 153Sm-EDTMP With Vaccine
Number analyzed (Participants) | 18 | 21
participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0

10. Secondary Outcome: Palliation: Pain at Baseline
Description: Subjective report of participant pain at baseline.This data reflects National Cancer Institute (NCI) patients only. This data was not systematically captured, so these results are based on subjective patient reports of improvement in pain on a scale of 1-10 post quadramet (samarium) as documented in the progress notes. 1-2 equals mild pain and 9-10 equals worst possible pain.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Arm A - EDTMP Alone | Arm B - 153Sm-EDTMP With Vaccine
Number analyzed (Participants) | 14 | 13
participants | 10 | 8

11. Secondary Outcome: Palliation: Improvement in Baseline Pain
Description: Subjective report of participant pain at baseline. This data reflects National Cancer Institute (NCI) patients only. This data was not systematically captured, so these results are based on subjective patient reports of improvement in pain on a scale of 1-10 post quadramet (samarium) as documented in the progress notes. 1-2 equals mild pain and 9-10 equals worst possible pain.
Time Frame: post quadramet (samarium)
Measure: Number; unit: participants
Arm/Group | Arm A - EDTMP Alone | Arm B - 153Sm-EDTMP With Vaccine
Number analyzed (Participants) | 10 | 8
participants | 6 | 5

ADVERSE EVENTS:
Arm/Group | Arm A -EDTMP Alone | Arm B - 153SmEDTMP With Vaccine
Serious Adverse Events (participants affected / at risk) | 5/21 | 5/22
Other Adverse Events (participants affected / at risk) | 19/21 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A -EDTMP Alone (N=21) | Arm B - 153SmEDTMP With Vaccine (N=22)
Anemia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (3) | 0 (0)
Pain (General disorders) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 1 (3)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Infections and infestations, Other, specify (Infections and infestations) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A -EDTMP Alone (N=21) | Arm B - 153SmEDTMP With Vaccine (N=22)
Alanine aminotransferase increased (Investigations) | 4 (4) | 0 (0)
Alkaline phosphatase increased (Investigations) | 9 (13) | 10 (15)
Anemia (Blood and lymphatic system disorders) | 12 (28) | 18 (45)
Anorexia (Metabolism and nutrition disorders) | 8 (8) | 8 (11)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 6 (8) | 6 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (2) | 0 (0) — absolute eosinophils decreased; neutrophils elevated
Blood bilirubin increased (Investigations) | 3 (3) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (12)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
CPK increased (Investigations) | 2 (2) | 0 (0)
Cardiac disorders - Other, (sinus tachycardia) (Cardiac disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (6) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 2 (4) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Edema: limbs (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 10 (13) | 12 (24)
Fever (General disorders) | 3 (3) | 3 (7)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Hematoma (Vascular disorders) | 2 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (3) | 2 (2)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 8 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (6) | 4 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (4) | 6 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (12) | 6 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (7) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 6 (7) | 1 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Hypotension (Vascular disorders) | 1 (3) | 1 (1)
INR increased (Investigations) | 1 (1) | 1 (1)
Investigations-Other, specify (Investigations) | 2 (2) | 2 (3) — bicarbonate serum low; troponin decreased
Lymphocyte count decreased (Investigations) | 11 (19) | 11 (21)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 (6) | 2 (3) — BUN (27); bicarbonate (22.8); creatinine (1.5); creatinine (2.3); creatinine decreased; total protein decreased; BUN 28; Elevated BUN; Low ALT
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder-Other, specify (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) — unsteady gait; jaw nodule
Nausea (Gastrointestinal disorders) | 8 (11) | 7 (8)
Nervous system disorders - Other, (sensory neuropathy) (Nervous system disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 8 (15) | 16 (43)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 6 (6) | 9 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 3 (3)
Platelet count decreased (Investigations) | 14 (29) | 19 (56)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 8 (12)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0) — trace bacteria in urine
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (5) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (6) | 4 (4)
Weight loss (Investigations) | 5 (6) | 5 (5)
White blood cell decreased (Investigations) | 14 (29) | 17 (49)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 4 (5)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 7 (9)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 4 (6)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 3 (3)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (3)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Infections and infestations, Other, specify (Infections and infestations) | 0 (0) | 1 (2) — infection skin Zoster right back
Injection site reaction (General disorders) | 0 (0) | 11 (34)

LIMITATIONS AND CAVEATS:
This study was stopped before full accrual(after about two-thirds of the subjects were enrolled) due to a significant decrease in enrollment despite making this a multicenter study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No